CLINICAL TRIAL: NCT01607242
Title: Study of Total Thyroidectomy Effect on Voice and Swallowing Function
Brief Title: Impact of Total Thyroidectomy on Voice and Swallowing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Jiannis Hajiioannou, ENT Consultant Lecturer University of Thessaly, University of Thessaly
Other Study IDs: thyro25
Record Dates: First submitted 2012-05-22; First posted 2012-05-30 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Thyroidectomy; Voice Alteration; Swallowing Alteration
Keywords: total thyroidectomy; voice handicap index; swallowing disorders; thyroid surgery; voice disorders
MeSH Terms: conditions — Dysphonia; Deglutition Disorders; Voice Disorders | interventions — Laryngoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients: patients undergoing total thyroidectomy
  Interventions: Other: Endoscopy of larynx; Other: Voice Handicap Index; Other: Swallowing Assesment

INTERVENTIONS:
Other: Endoscopy of larynx — Endoscopic Laryngeal mobility assessment
Other: Voice Handicap Index — Subjective Evaluation of Voice disorders
Other: Swallowing Assesment — Swallowing function questionnaire

SUMMARY:
Purpose of this study is to evaluate the outcome of total thyroidectomy on vocal and swallowing function.

DETAILED DESCRIPTION:
Voice and swallowing alterations are frequently reported after thyroidectomy, even in the absence of nerve injury. These impair quality of life.

Purpose of this study is to evaluate the outcome of total thyroidectomy on vocal and swallowing function.

Patients will be assessed using the Greek- version of Voice Handicap Index (VHI) and a questionnaire developed by the authors regarding swallowing symptoms.

Furthermore they will undergo flexible laryngoscopy for evaluation of laryngeal mobility.

ELIGIBILITY:
Inclusion Criteria:

* All patients submitted to total thyroidectomy during the study period

Exclusion Criteria:

* Previous thyroid/ neck surgery
* Documented voice disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing total thyroidectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-03

PRIMARY OUTCOMES:
Subjective voice evaluation | 1 Day preoperatively
  Greek- version of Voice Handicap Index (VHI)
Subjective voice evaluation | 1 week postoperatively
  Greek- version of Voice Handicap Index (VHI)
Subjective Voice Evaluation | 1 month postoperatively
  Greek- version of Voice Handicap Index (VHI)

SECONDARY OUTCOMES:
Swallowing evaluation | 1 day preoperatively
  questionnaire on swallowing symptoms
Swallowing evaluation | 1 week postoperatively
  questionnaire on swallowing symptoms
Swallowing evaluation | 1 month postoperatively
  questionnaire on swallowing symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Bizakis, Professor, Study Chair — University of Thessaly; Jiannis Hajiioannou, Lecturer, Principal Investigator — University of Thessaly; Evangelos Athanasiou, As Professor, Study Chair — University of Thessaly; Dimitrios Zacharoulis, As Professor, Study Director — University of Thessaly; Eleni Sioka, MD, Study Director — University of Thessaly; Vassilios Lachanas, MD, Study Director — University of Thessaly
Locations (1):
- University Hospital of Larissa, Larissa, Greece

REFERENCES:
- [Background] Helidoni ME, Murry T, Moschandreas J, Lionis C, Printza A, Velegrakis GA. Cross-cultural adaptation and validation of the voice handicap index into Greek. J Voice. 2010 Mar;24(2):221-7. doi: 10.1016/j.jvoice.2008.06.005. Epub 2008 Aug 26. PMID 18752925
- [Background] de Pedro Netto I, Fae A, Vartanian JG, Barros AP, Correia LM, Toledo RN, Testa JR, Nishimoto IN, Kowalski LP, Carrara-de Angelis E. Voice and vocal self-assessment after thyroidectomy. Head Neck. 2006 Dec;28(12):1106-14. doi: 10.1002/hed.20480. PMID 16933312
- [Background] Lombardi CP, Raffaelli M, D'alatri L, De Crea C, Marchese MR, Maccora D, Paludetti G, Bellantone R. Video-assisted thyroidectomy significantly reduces the risk of early postthyroidectomy voice and swallowing symptoms. World J Surg. 2008 May;32(5):693-700. doi: 10.1007/s00268-007-9443-2. PMID 18259807